CLINICAL TRIAL: NCT05469295
Title: A Prospective, Randomized, Single-blinded, Sham Device Controlled, Parallel Treatment Grouped, Multi-center, Exploratory Clinical Trial to Evaluate Improvement of Cervical Lordosis and Safety of CGM MB-1701 in Subjects With Cervical Kyphosis and Posterior Neck Pain.
Brief Title: CETIC-I (CEra Traction Improves Cervical Kyphosis -I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceragem Clinical Inc. (Industry)
Responsible Party: Sponsor
Organization: Ceragem Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRG_MV6_P03
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cervical Kyphosis; Cervical Lordosis; Kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM_MB_1701 treatment (Experimental): Subjects will be treated with the study device for about 36 minutes.
  Interventions: Device: CGM MB-1701 device treatment
- Sham (CGM MB1701C) treament (Sham Comparator): Subjects will be treated with the Sham device for about 36 minutes.
  Interventions: Device: CGM MB-1701 Sham device treatment

INTERVENTIONS:
Device: CGM MB-1701 device treatment — This is a pre-approved motorized traction device.
  Arms: CGM_MB_1701 treatment
Device: CGM MB-1701 Sham device treatment — It is manufactured in the same way as the test device and the operation pattern. However, the actual effect of the massage is minimized.
  Arms: Sham (CGM MB1701C) treament

SUMMARY:
The study is a Prospective, Randomized, Single-blinded, Sham device controlled, Parallel Treatment Grouped, Multi-center, Exploratory Clinical Trial to Evaluate Improvement of Cervical Lordosis and Safety of CGM MB-1701 (Spinal warm massage device, Ceragem Master V6) in Subjects with Cervical Kyphosis and Posterior Neck Pain.

DETAILED DESCRIPTION:
The Cervical Kyphosis are also commonly referred to as "turtle neck syndrome." It refers to the deformation of the neck bone into an inverted C-shape due to abnormalities or degenerative changes, and it is named to mean that the neck is bent like a turtle.

This device, Ceragem Master V6 (CGM MB-1701), has been certified as a combination of a personal warmer that can be used to relieve muscle pain by applying constant heat to the human body and a medical vibrator of a device that applies physical energy (vibration, shock, pressure, etc.). Also, the device got approval for use with intermittent pneumatic compression and electrically-powered orthopedics traction.

The primary purpose of this clinical trial is to confirm the temporary cervical lordosis angle improvement (height) in subjects with cervical kyphosis through the combined function of the test device.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects who have voluntarily decided to participate and agreed in writing after being briefed on the characteristics of this clinical trial and medical device
2. Subjects with cervical kyphosis angle between cervical lordosis 20 degrees and cervical kyphosis 5 degrees.
3. BMI betweeen 18.5 and 30
4. Chronic neck pain NRS 4 or higher lasting more than 3 months

Exclusion Criteria:

1. Secondary spondylosis
2. A tumor of the spine
3. Inflammatory spondylitis
4. Myelopathy
5. Multiple adjacent radiculopathies and others

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Mean change of cervical lordosis | up to 16 weeks
  Mean change of cervical lordosis using posterior tangent method of Harrison measured by cervical lateral radiography at EOT (End of Trial) compared to baseline.

SECONDARY OUTCOMES:
Change of cervical lordosis at 2nd interim analysis | up to 16 weeks
  Change of the cervical lordosis (posterior tangent method of Harrison) measured by cervical lateral radiography at the 2nd interim visit compared to baseline.
Cervical vestibular angle increase more than 10 degrees | up to 16 weeks
  The fraction of subjects whose cervical vestibular angle measured by the posterior tangent method of Harrison at each time of evaluation increased by more than 10 degrees compared to the baseline
Anteroposterior (T1) slope average change | up to 16 weeks
  Average change in cervical anteroposterior (T1) slope measured by cervical lateral radiography at each evaluation compare to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yong Il Shin, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No